CLINICAL TRIAL: NCT05306912
Title: Molecular Analysis of Endoscopic Cytology Samples Supernatant in Pulmonary Nodules (Cancer Or Benign Endoscopy) (KOBE)
Brief Title: Molecular Analysis of Endoscopic Cytology Samples Supernatant in Pulmonary Nodules
Acronym: KOBE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC31/20/0446; ID-RCB 2021-A01024-37 (Other: ANSM); ARI 20-0446 (Other Grant/Funding Number: University Hospital, Toulouse)
Record Dates: First submitted 2022-03-01; First posted 2022-04-01 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Lung Cancer; Lung; Node
Keywords: Circulating free DNA; Methylation; Lung cancer; screening; lung nodule; radial EBUS; endobronchial ultrasound
MeSH Terms: conditions — Lung Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- blood sampling (Experimental): blood sample (2 tubes of 7.5 mL of blood = 15 mL) during the preoperative check-up on the day of the ultrasound-bronchoscopy in order to compare the sensitivity of the analysis of free circulating DNA present in the supernatant of pulmonary nodules less than 20 mm samples taken under ultrasound-bronchoscopy to that present in the plasma
  Interventions: Biological: Blood samples

INTERVENTIONS:
Biological: Blood samples — Patients will be taken from an additional blood sample (2 tubes of 7.5 mL of blood = 15 mL) during the preoperative check-up on the day of the ultrasound-bronchoscopy in order to compare the sensitivity of the analysis of free circulating DNA present in the supernatant of pulmonary nodules less than 20 mm samples taken under ultrasound-bronchoscopy to that present in the plasma.

SUMMARY:
Lung cancer screening is based on low dose CT scan (LDCT), a highly sensitive but poorly specific tool.

Complementary specific approaches are thus strongly needed, among which cell-free DNA (cfDNA) genotyping has been proven highly specific but of low sensitivity (25 to 50% for stage I diseases) due to inconstant tumor shed. Tumor biopsy is thus often required and radial endobronchial ultrasound (rEBUS) bronchoscopy is a minimally invasive approach (<3% complications) but of limited sensitivity in cases of nodules < 20 mm.

The investigators hypothesized that methylation analysis on cfDNA floating in supernatant derived from rEBUS specimens could improve rEBUS sensitivity

DETAILED DESCRIPTION:
Tumor biopsy is often required to characterize indeterminate nodules. Radial endobronchial ultrasound (rEBUS) bronchoscopy is often used due to a low rate of complications but its sensitivity is limited for small nodules.

The investigators hypothesized that methylation analysis on cfDNA floating in supernatant derived from rEBUS specimens could improve rEBUS sensitivity.

The primary outcome of this pilot, diagnostic validation, monocentric study is the sensitivity of targeted (9 genes panel) methylation analysis on supernatant cfDNA to detect a malignant nodule.

Secondary outcomes include the comparison of supernatant to pathology and plasma cfDNA methylation analysis.

Specificity, negative predictive value (NPV), positive predictive value (PPV) of targeted (9 genes panel) methylation analysis on supernatant cfDNA to detect a malignant nodule will be analyzed.

60 patients planned for a rEBUS bronchoscopy for one, two or three < 20 mm nodule, without mediastinal or extra thoracic lesions (cT1N0M0) will be included.

The day of the rEBUS bronchoscopy, 2 7.5 mL blood samples are collected. rEBUS samples' supernatant, usually discarded, is saved.

Cell free DNA is extracted from these biological specimens at the Laboratory of Oncological Medical Biology (LBMO) in Toulouse University Cancer Institute and tested for methylation (targeted analysis on 9 genes).

The patients will be followed for one year to obtain a final diagnosis and correlate it with tissue, nodule supernatant and plasma methylation analyses.

ELIGIBILITY:
Inclusion Criteria:

* rEBUS bronchoscopy planned for one, two or three ≤ 20 mm nodule
* World Health Organization (WHO) Performance status 0-3
* Informed signed consent
* Patient affiliated or beneficiary of a social security scheme (Social Security or Universal Medical Coverage).

Exclusion Criteria:

* Lung cancer diagnosed before the date of the procedure
* Lung cancer strongly suspected due to mediastinal or extra thoracic lesions
* Patient under State Medical Assistance
* Patient deprived of liberty on administrative or judicial decision, or patient under guardianship, curators or safeguard of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-04-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of targeted (9 genes panel) methylation analysis on supernatant cfDNA to detect a malignant nodule will be evaluated. | 1st day (D0) of patients' inclusion, on morning of their ultrasound-bronchoscopy
  Promoter methylation rates of the 9 targeted genes in the free circulating DNA of the endoscopic samples supernatant is obtained by quantitative Polymerase Chain Reaction (PCR) of bisulfite-treated DNA fragments from the cytological samples supernatant after DNA concentration and separation by size at the Centre of Cancer Research of Toulouse (CRCT).
  These analyses will be performed blinded to the clinical data and the histopathology result of the lung nodule.

SECONDARY OUTCOMES:
Comparison of supernatant to pathology and plasma cfDNA methylation analysis. Specificity, negative predictive value (NPV), positive predictive value (PPV) of targeted (9 genes panel) methylation analysis on supernatant cfDNA to detect a malignant nodule | 1st day (D0) of patients' inclusion, on morning of their ultrasound-bronchoscopy
  Methylation profiles of free circulating DNA from plasma obtained after centrifugation of blood samples will be obtained by the same method as described for analysis of cytopunction's supernatant methylation profile.
  These analyses will be performed blinded to the clinical data and the histopathology result of the lung nodule.

CONTACTS AND LOCATIONS:
Overall Officials: Valentin HELUAIN, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Toulouse University Hospital, Toulouse, Occitanie, France

IPD SHARING:
Plan to Share IPD: No